CLINICAL TRIAL: NCT06020287
Title: The Early Therapeutic Efficacy of The Robot-Assisted Laparoscopic Radical Prostatectomy Combined Anterior and Posterior Approach: A Single-Center Retrospective Cohort Study
Brief Title: The Robot-Assisted Laparoscopic Radical Prostatectomy Combined Anterior and Posterior Approach
Status: Completed | Type: Observational
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Fan Feng, Attending Doctor, Nanjing University School of Medicine
Other Study IDs: NanjingUSM202388
Record Dates: First submitted 2023-08-08; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Prostatectomy; Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AP-RARP: the robot-assisted laparoscopic radical prostatectomy combined anterior and posterior approach
  Interventions: Procedure: the robot-assisted laparoscopic radical prostatectomy
- RS-RARP: the robot-assisted laparoscopic radical prostatectomy with the Retzius-sparing approach
  Interventions: Procedure: the robot-assisted laparoscopic radical prostatectomy
- anterior-RARP: he robot-assisted laparoscopic radical prostatectomy with anterior approach
  Interventions: Procedure: the robot-assisted laparoscopic radical prostatectomy

INTERVENTIONS:
Procedure: the robot-assisted laparoscopic radical prostatectomy — We collect medical data of 233 patients with clinically localized prostate cancer who underwent AP-RARP, RS-RARP or anterior-RARP. Perioperative outcomes, including operation time, intraoperative blood loss, intraoperative and postoperative transfusion, postoperative infection, and anastomotic leakage, were compared among the three groups. The postoperative continence rates and PSM rates were also compared.

SUMMARY:
The goal of this observational study was to compare the perioperative outcomes, postoperative urinary control rates and positive surgical margin (PSM) rates of the robot-assisted laparoscopic radical prostatectomy combined anterior and posterior approach (AP-RARP) with the Retzius-sparing approach (RS-RARP) and anterior approach (anterior-RARP) in the treatment of prostate cancer. The main question it aims to answer was:

• The early therapeutic efficacy of the robot-assisted laparoscopic radical prostatectomy combined anterior and posterior approach

Participants has been underwent:

* AP-RARP
* RS-RARP
* anterior-RARP Researchers compared the three groups to see if AP-RARP combines the advantages of anterior and posterior RARP and is a feasible surgical option for the treatment of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed with prostate cancer by prostate biopsy
* underwent robot-assisted laparoscopic surgery
* the surgery performed by Weidong Gan
* the extended pelvic lymphadenectomy (PLA) is performed on patients with high-risk prostate cancer (PSA≥20 ng/ml or Grade Group 4-5 or clinical stage ≥T2c) and those considered to have a possibility of lymph node metastasis based on imaging evaluation.

Exclusion Criteria:

* Patients with a clinical and pathological TNM stage ≥T3b and N1
* patients with distant metastasis
* urinary incontinence before surgery
* received neoadjuvant therapy before surgery

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The clinical data of 233 patients treated between September 2020 and May 2022 at Nanjing Drum Tower Hospital were retrospectively analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
urinary continence | 0-6 month after surgery
  was defined as using 0-1 pad a day
positive surgical margin | 2 weeks after surgery
  observed whether the tissue cutting in surgery has tumor cell in surgical margin by pathologist

SECONDARY OUTCOMES:
operating time | the day of the surgery
  The start time of the operation refers to the time of incision of the skin at the surgical site. The end time of surgery refers to the time when the skin is sutured.
intraoperative blood loss | the day of the surgery
  Intraoperative bleeding was defined as the sum of blood content in blood gauze, blood content in negative pressure suction bottle and blood clot volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided